CLINICAL TRIAL: NCT05388149
Title: Kadcyla And Neratinib for Interception of HER2+ Breast Cancer With Molecular Residual Disease
Status: Recruiting | Phase: Phase 2 | Type: Interventional
Sponsor: University Health Network, Toronto (Other)
Responsible Party: Sponsor
Allocation: Not Applicable | Model: Single Group | Masking: None | Purpose: Treatment
Other Study IDs: 22-5307; KAN-HER2 MRD (Other: UHN)
Record Dates: First submitted 2022-05-18; First posted 2022-05-24 (Actual); Last update posted 2025-01-31 (Actual); Status verified 2025-01

CONDITIONS: Breast Cancer; HER2-positive Breast Cancer
MeSH Terms: conditions — Breast Neoplasms | interventions — neratinib

STUDY DESIGN:
Oversight: Data Monitoring Committee: Yes | FDA-regulated Drug: No | FDA-regulated Device: No

ARMS (1):
- Neratinib Arm (Experimental): Standard T-DM1 (3.6mg/kg) IV infusion every 3 weeks administered with Neratinib (160 mg) orally once daily up to 1 year.
  Interventions: Drug: Neratinib

INTERVENTIONS:
Drug: Neratinib — Neratinib administered as 40mg tablets
  Other Names: NERLYNX

SUMMARY:
This is a Phase 2 study for patients with resected Stage I-III HER2+ breast cancer with detected molecular residual disease (MRD+) following standard neoadjuvant and locoregional therapy delivered with curative intent. In this study Patients will be treated with neratinib in addition to their standard T-DM1 adjuvant therapy. Neratinib will be administered orally at a dose of 160 mg daily for up to 12 months, or until the time of clinical recurrence, discontinuation due to toxicity, or withdrawal of consent. This study will have two stages, stage 1 would enroll up to 8 participants to clear the Minimal Residual Disease (MRD) and Stage 2 will enroll up to 5 participants. The purpose of this study is to determine if this study population would have a better outcome from adding neratinib to their standard T-DM1 adjuvant therapy.

ELIGIBILITY:
Inclusion Criteria:

1. Male or female patients ≥ 18 years of age with histologically confirmed, resected HER2 positive stage I-III breast cancer, with residual invasive disease following prior neoadjuvant trastuzumab (+/- pertuzumab)-based chemotherapy.
2. Receiving adjuvant T-DM1, with evidence of MRD (positive test by Inivata RaDaR) after receiving 2-6 cycles of T-DM1
3. No contraindications to T-DM1 or neratinib
4. No clinical or radiographic evidence of recurrent or metastatic disease
5. Previous Therapy requirements:

   * Received 2-6 cycles of trastuzumab-DM1 in the adjuvant setting
   * Received min of 12 weeks of endocrine therapy (ER+ patients)
   * Adjuvant radiation permitted (minimum 14-day washout required)
   * No prior neratinib or other HER2 tyrosine kinase inhibitor
6. ECOG performance status 0-1.
7. Patient must have adequate organ function
8. WOCBP must have a negative serum [beta] HCG test result.
9. WOCBP must agree to use highly effective contraception
10. Male participants must agree to use highly effective contraception
11. Subject is willing and able to comply with the protocol for the duration of the study including undergoing treatment and scheduled visits and examinations including follow up.
12. Signed informed consent

Exclusion Criteria:

1. Prior therapy with any HER2 tyrosine kinase inhibitor
2. Clinical or radiographic evidence of suspected or confirmed metastatic disease.
3. Previous or concurrent malignancy within 3 years of study entry, with exceptions
4. Impaired cardiovascular function or clinically significant cardiovascular diseases
5. Known positive serology for HIV that is not currently controlled with anti-retroviral therapy,
6. Has a known history of or is positive for active hepatitis B (defined as hepatitis B surface antigen [HBsAg] reactive) or hepatitis C (defined as HCV RNA [qualitative] is detected). HBV DNA must be undetectable and HBsAg negative at Screening Visit. Participants who have had definitive treatment for HCV are permitted if HCV RNA is undetectable at Screening Visit.
7. Impaired gastrointestinal function or disease that may significantly alter the absorption of neratinib
8. Medical, psychiatric, cognitive, or other conditions that may compromise the patient's ability to understand the patient information, give informed consent, comply with the study protocol, or complete the study.

Min Age: 18 Years | Sex: All | Healthy Volunteers: No
Age Groups: Adult, Older Adult
Enrollment: 15 (Estimated)
Dates: Start 2022-12-06 (Actual); Primary Completion 2026-07 (Estimated); Study Completion 2026-07 (Estimated)

PRIMARY OUTCOMES:
Clearance of ctDNA with the addition of neratinib to trastuzumab-DM1 in patients with MRD detectable by the RaDaR assay, following standard neoadjuvant therapy, surgery, and initiation of T-DM1 | At week 12

SECONDARY OUTCOMES:
Clinical outcomes for MRD+ patients treated with escalated strategy, including invasive breast cancer-free survival (IBCFS) measured by Invasive Breast Cancer-Free Survival and Distant Metastasis Free Survival | Up to 3 years
Toxicities of the combination of neratinib and trastuzumab-DM1 in the study population measured by CTCAE 5.0 | Up to 3 years
Characterize dynamic changes and kinetics in ctDNA MRD+ for enrolled patients measured by ctDNA MRD Detection by RaDaR assay | Up to 3 years

CONTACTS AND LOCATIONS:
Locations (1):
- University Health Network: Princess Margaret Cancer Centre, Toronto, Ontario, Canada

IPD SHARING:
Plan to Share IPD: No